CLINICAL TRIAL: NCT03184038
Title: Neurocognition in Patients With Multiple Brain Metastases Treated With Radiosurgery: A Phase II Study
Brief Title: Neurocognition in Patients With Multiple Brain Metastases Treated With Radiosurgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16D.651; JT 9331 (Other: JeffTrial Number)
Record Dates: First submitted 2017-04-05; First posted 2017-06-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Mental Status and Dementia Tests; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (SRS/SBRT, neurocognitive testing) (Experimental): Patients undergo SRS on day 1 or SBRT for 3 fractions over days 1-7 and undergo neurocognitive testing at baseline, 4, and 12 months after undergoing SRS or SBRT.
  Interventions: Procedure: Cognitive Assessment; Radiation: Stereotactic Radiosurgery; Radiation: Stereotactic Body Radiation Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Cognitive Assessment — Undergo assessment of neurocognitive function
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT; SABR; Stereotactic Ablative Body Radiation Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the neurological function in patients with multiple brain metastases undergoing stereotactic radiosurgery (SRS) or stereotactic body radiation therapy (SBRT). Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Assessment of neurocognitive function may help show that SRS preserves neurological function in patients with multiple brain metastases better than SBRT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assessment of neurocognitive function at months 4.

SECONDARY OBJECTIVES:

I. Assessment of neurocognitive function at months 4 and 12 as measured by neurocognitive decline on a battery of tests.

II. Assessment of symptom burden, as measured by the M.D. Anderson Symptom Inventory- Brain Tumor Module (MDASI-BT).

III. Assessment of quality adjusted survival and health outcomes using the European Quality of Life Five Dimension Five Level scale questionnaire (EQ-5D-5L).

IV. Assessment of local control, in brain control. V. Assessment of progression free survival (PFS), and overall survival (OS). VI. Assessment of side effects and toxicities.

OUTLINE:

Patients undergo SRS on day 1 or SBRT for 3 fractions over days 1-7 and undergo neurocognitive testing at baseline, 4, and 12 months after undergoing SRS or SBRT.

After completion of study, patients are followed up at 2, 4, 6, 8, 10, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven solid tumor malignancy (except for small cell lung cancer [SCLC], germ cell tumor)
* Karnofsky performance status >= 60
* 1 to 10 brain metastases (mets) (no more than two lesions and/or cavities >= 3 cm in maximum diameter)
* Maximum diameter of brain metastasis or resection cavity is 6 cm
* Serum creatinine =< 3 mg/dL and creatinine clearance >= 30 ml/min
* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up; patients must be willing to complete neurocognitive assessments at pre-specified time points outlined in the protocol
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test documented within 21 days prior to registration
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 4 months after last dose
* Patient able to provide his/her own written informed consent and speak English

Exclusion Criteria:

* Patient with diagnosis of glioma, or other World Health Organization (WHO) grade II - IV primary brain tumor
* Prior brain surgery =< 14 days prior to enrollment
* Planned chemotherapy during radiosurgery
* Leptomeningeal metastases
* Intractable seizures while on adequate anticonvulsant therapy-more than 1 seizure per week for the past 2 months
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive function as measured by neurocognitive decline on a battery of tests | At 4 months
  The proportion of patients with neurocognitive decline at 4 months post stereotactic radiosurgery (SRS) treatment in each group will be estimated using the sample proportion with the corresponding two-sided 95% confidence interval. The determination of neurocognitive decline will be based on a battery of tests: Hopkins Verbal Learning Test-Revised (HVLT-R) for Total Recall, Delayed Recall, and Delayed Recognition, Controlled Oral Word Association (COWA), and the Trail Making Test (TMT) Parts A and B. The operative definition for neurocognitive decline in this study will be decline on at least one of these measures.

SECONDARY OUTCOMES:
Change in neurocognitive function as measured by neurocognitive decline on a battery of tests conducted by the primary investigator or a trained member of the clinical team | Baseline to up to 12 months
  Each patient will serve as his or her own control, and the relative decline in HVLT-R scores from baseline to pre-specified post-treatment internals will be defined as follows: ΔHVLTi = (HVLTB - HVLTF) ÷ HVLTB, where B = baseline and F = follow-up. A positive change indicates a decline in function. Comparison of HVLT-R DR results between control and different time points will be tested using the one-side Wilcoxon signed rank test with significance level of .05. The repeated measures of each neurocognitive test (HVLT-R, COWA, and TMT) and the health-related quality of life (HR-QOL) scale at 2, 4, 6, and 12 months will be analyzed using a linear mixed effects model. The dichotomous indicator of neurocognitive decline based on this battery of tests at 2, 4, 6, and 12 months will be analyzed using a repeated measures logistic regression model.
Change in symptom burden as measured by the MD Anderson Symptom Inventory- Brain Tumor Module (MDASI-BT) | Baseline to up to 12 months
  Four subscales (symptom severity, symptom interference, neurologic factor, and cognitive factor score) as well as certain individual items (fatigue, neurologic factor items, and cognitive factor items) of the MDASI-BT will be analyzed. For discrete time point analyses, the change from baseline to each follow-up time point (2, 4, 6, and 12 months from the start of treatment) will be calculated and compared between treatment arms using a t-test or Wilcoxon-Mann-Whitney test, depending on the normality of the data.
Quality adjusted survival and health outcomes as measured by the European Quality of Life Five Dimension Five Level scale questionnaire (EQ-5D-5L) | Up to 12 months
  The Z-test will be used to test the hypothesis that the health outcomes in the 2 treatment groups is the same at different time points after initiation of treatment with a significance level of 0.05 and a 2-sided test.
Local control as measured by magnetic resonance imaging | Up to 12 months
  Will be measured by magnetic resonance imaging.
Progression free survival (PFS) | Up to 12 months
  Each group will be evaluated using the Kaplan-Meier method.
Overall survival (OS) | Up to 12 months
  Each group will be evaluated using the Kaplan-Meier method.
Incidence of adverse events graded according to the Common Terminology Criteria for Adverse Events version 5.0 | Up to 30 days after SRS
  Descriptive analysis will be performed on the acute toxicity data. All estimates of rates (e.g., discontinuation rate and rates of other toxicities) will be presented with corresponding confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (2):
- United States (2):
  - Jefferson Health New Jersey, Sewell, New Jersey
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/